CLINICAL TRIAL: NCT02506452
Title: Evaluation of Biovance, a Dehydrated Decellularized Human Amniotic Membrane Allograft, in Diabetic Foot Ulcers
Brief Title: Postmarket Study to Evaluate Biovance® in Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliqua BioMedical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALQ.BIO.2015.01
Record Dates: First submitted 2015-07-21; First posted 2015-07-23 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded wound core lab
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biovance® (Active Comparator): Application of Biovance® for up to 12 weeks or until wound closure, whichever is sooner. Non-active moist wound treatment, debridement as needed, off-loading device
  Interventions: Other: Biovance®; Other: Standard of Care, Diabetic Foot Ulcers
- Standard of Care, Diabetic Foot Ulcers (Active Comparator): Non-active moist wound treatment, debridement as needed, off-loading device
  Interventions: Other: Standard of Care, Diabetic Foot Ulcers

INTERVENTIONS:
Other: Biovance® — Application of Biovance® for up to 12 weeks or until wound closure, whichever is sooner. Non-active moist wound treatment, debridement as needed, off-loading
  Arms: Biovance®
Other: Standard of Care, Diabetic Foot Ulcers — Non-active moist wound treatment, debridement as needed, off-loading for up to 12 weeks or until wound closure, whichever is sooner

SUMMARY:
The purpose of this study is to compare the wound closure outcomes of subjects receiving diabetic foot ulcer treatment with and without the use of Biovance®.

ELIGIBILITY:
Inclusion Criteria:

* The subject has:

  1. been diagnosed with Diabetes Mellitus (insulin or non-insulin dependent) and peripheral neuropathy (loss of protective sensation) in affected foot
  2. a HbA1c of less than 10% assessed within last 12 weeks
  3. a full-thickness diabetic neuropathic foot ulcer that is free from tunnels/sinus tracks, necrotic tissue, exposed bone and/or tendon, and osteomyelitis post debridement (Wagner 1 or 2; Appendix I)
  4. one (target) diabetic neuropathic foot ulcer of less than 12 months duration that has an area that measures ≥ 1.5 and ≤ 10 cm2 post debridement (max length x max width) at screening that is on any surface and part of the foot (fore-, mid- or hind-foot) with an etiology related to loss of protective sensation in that foot.
  5. a target ulcer that closed <30% during the 2 week run-in period (2 weeks management with SOC following signature of informed consent prior to potential randomization)
  6. sufficient arterial supply to affected foot tested within the past 60 days

Exclusion Criteria:

* The subject has:

  1. ulcers of non-diabetic etiology on the study foot
  2. a target ulcer clinically infected or has underlying osteomyelitis at time of study treatment initiation
  3. clinical evidence of gangrene on any part of the affected foot
  4. a target ulcer with exposed bone or tendon
  5. any malignancy or a neoplasm at the target ulcer site
  6. active Charcot Foot or Charcot Foot that is unable to be offloaded (stable, non-active Charcot deformity that is able to be offloaded is acceptable)
  7. more than 3 ulcers on the study foot, including the target ulcer, and all other ulcers must be at least 3 cm removed from the target ulcer
  8. any significant comorbid disease that may interfere with wound healing
  9. received chemotherapy, radiotherapy, immunosuppressant or corticosteroid (greater than 10 mg prednisone-equivalent per day) within the past 30 days.
  10. had the diabetic foot ulcer treated with an experimental drug/biologic/device, or a live-cell therapy (experimental or marketed), or active moist wound healing therapy within 30 days of randomization day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Wound closure observed at up to 12 weeks following baseline visit defined as 100% re-epithelialization without drainage confirmed at 2 weeks following initial observation of closure. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Institute of Advanced Wound Healing, Montgomery, Alabama
  - Banner Health, Phoenix, Arizona
  - Limb Preservation Platform, Fresno, California
  - Southern California Institute for Research and Education (VA), Long Beach, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Georgetown University, Washington D.C., District of Columbia
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - Foot and Ankle Center at Coordinated Health, Bethlehem, Pennsylvania
  - University of Tennessee Health Sciences Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No